CLINICAL TRIAL: NCT03275935
Title: Evaluation of Inhalation Technique in Patients With Chronic Obstructive Pulmonary Disease (COPD), Asthma or Asthma-COPD Overlap Syndrome(ACOS) Using a Dry Powder Device at Chest Clinic in Dhulikhel Hospital
Brief Title: Evaluation of Inhalation Technique in Patients With COPD, Asthma or ACOS Using a Dry Powder Device (DPI)
Status: Completed | Type: Observational
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Sudeep Shrestha, Lecturer, CardioPulmonology Unit, Department of Internal Medicine, Kathmandu University School of Medical Sciences
Other Study IDs: 73/17
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: COPD Asthma; Asthma-COPD Overlap Syndrome; Inhalation
Keywords: ACOS; Asthma; COPD; inhalation technique
MeSH Terms: conditions — Asthma-Chronic Obstructive Pulmonary Disease Overlap Syndrome; Respiratory Aspiration; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Training Arm: Patients that were given training in regards to proper inhalation technique of Rotahalers

SUMMARY:
This study analyzes the prevalence of patients using inhalation devices via incorrect technique and access the adherence of patients to correct inhalation technique when taught along with their subjective improvement of symptoms.

DETAILED DESCRIPTION:
This is a one group pretest- posttest design conducted in all patients presenting in Chest clinic of Dhulikhel Hospital-Kathmandu University Hospital, Nepal from March 2017 to May 2017. Patients diagnosed of having COPD, Asthma or Asthma-COPD Overlap Syndrome (ACOS) and were under inhalation bronchodilators in the form of Dry Powder Device via Rotahaler were included. Enrolled patients are assessed for inhalation technique compliance at their routine medical (pre-training) visits by physician. The use of inhaler device is evaluated in a practical manner by asking the patients to demonstrate their inhalation technique. After the assessment, instructions and training are given until they can use the device correctly. One month later (post-training), all patients are re-evaluated in regards to inhalation technique and subjective improvement of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years,
* Diagnosed of having of asthma or COPD or ACOS
* Using dry powder inhaler therapy with Rotahaler

Exclusion Criteria:

* Use of inhaler devices other than Rotahaler
* Newly started on dry powdered inhalational therapy or patients who had recently received face-to-face training program on inhalation technique within the past one month
* Patients in acute exacerbation
* Patients failing to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to Chest Clinic of Dhulikhel hospital, who were diagnosed of having either COPD, Asthma or Asthma-COPD Overlap Syndrome and are currently under inhalational bronchodilators in the form of Dry Powder Device (DPIs)
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in 'Inhalation Scores" After a month from Baseline | After a month
  An observation checklist measuring essential steps required for adequate drug delivery for Rotahaler was developed. The number of required steps are seven and the correctness of the seven-step inhalation technique was measured by giving a score 0 for incorrect action and 1 for correct action. Each of the seven steps were scored 1 or 0, giving a total score of 0-7. After assessment, instructions were given with demonstrations regarding the correct use of Rotahaler. One month later (post-training visit), all patients were re-evaluated

SECONDARY OUTCOMES:
Prevalance COPD, Asthma and Asthma COPD Overlap Syndrome inpatients visiting Chest Clinic of Dhulikhel Hospital- Kathmandu University Hospital. | 3 months
  Calculating the prevalence of the three medical conditions in Chest clinic of Dhulikhel Hospital
Associated Factors for Incorrect Inhalation Technique | 3 months
  The potential associated factors for an incorrect inhalation technique to be calculated via univariable logistic regression analysis
Prevalence of patients using the inhalation devices via incorrect technique | At pretraining
  An observation checklist measuring essential steps required for adequate drug delivery for Rotahaler was developed. The number of required steps are seven and the correctness of the seven-step inhalation technique was measured by giving a score 0 for incorrect action and 1 for correct action. Each of the seven steps were scored 1 or 0, giving a total score of 0-7.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sudeep Shrestha, MD, MRCP(UK), Principal Investigator — Dhulikhel Hospital- Kathmandu University Hospital
Locations (1):
- Dhulikhel Hospital- Kathmandu University Hospital, Dhulikhel, Nepal

IPD SHARING:
Plan to Share IPD: Undecided